CLINICAL TRIAL: NCT01995955
Title: The Proposed Study is to Validate a New Non-invasive Imaging Technique for Evaluation of Cardiac Microciculation in Coronary Artery Disease With a Comparison With Validated Technique Invasive, Which is Measure of Index of Myocardial Resistance
Brief Title: Evaluation of Coronary Microvascular Dysfunction (EVACORY)
Acronym: EVACORY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A00986-37
Record Dates: First submitted 2012-11-27; First posted 2013-11-27 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Microvascular Dysfunction; coronary artery disease; index of myocardial resistance
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- a new non-invasive imaging technique (Experimental): a new non-invasive imaging technique for evaluation of cardiac microciculation in coronary artery disease
  Interventions: Procedure: a new non-invasive imaging technique

INTERVENTIONS:
Procedure: a new non-invasive imaging technique — a new non-invasive imaging technique for evaluation of cardiac microciculation in coronary artery disease

SUMMARY:
The proposed study is to validate a new non-invasive imaging technique for evaluation of cardiac microciculation in coronary artery disease with a comparison with validated technique invasive, which is measure of index of myocardial resistance.

DETAILED DESCRIPTION:
Coronary microvascular dysfunction is closely associated with coronary artery disease, it is an independent risk factor and predicts future coronary events or clinically manifest disease up to 10 years later.

Index of microcirculatory resistance (IMR) is a validated method to Assessment of the Coronary Microcirculation but this is an invasive technique.

In this study, we use a new mathematic technique from homogeneity analysis to provide precise, objective, automated quantification of perfusion heterogeneity at stress with new camera CZT SPECT. We compare the results with those of the measurement of IMR.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina
* Cadmium-zinc-telluride gamma camera SPECT
* Coronarography

Exclusion Criteria:

* Pregnant woman
* Patient with terminal illness,
* Terminal Renal failure
* Allergy to iodine
* Contraindications for adenosine: Asthmatic patients, Second- or third-degree AV block without a pacemaker or sick sinus syndrome, Systolic blood pressure less than 90mm Hg, Recent use of dipyridamole or dipyridamole-containing medications, Methyl xanthenes such as aminophylline caffeine or theobromine block the effect of adenosine and should be held for at least 12 hours prior to the test, Known hypersensitivity to adenosine, Unstable acute myocardial infarction or acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-06-24 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
coronary microcirculation | day 0 (inclusion)
  IMR was measured with commercially available software (St Jude Medical Systems) and thermodilution technique on a non-ischemic artery SPECT. Injections of 3 mL of room-temperature saline were made down the coronary artery, and the resting mean transit time (Tmn) was measured. CFR was calculated as resting Tmn divided by hyperemic Tmn. FFR was calculated by the ratio of Pd/Pa at maximal hyperemia.IMR was defined as distal coronary pressure multiplied by the hyperemic mean transit time (mm Hg • seconds, or units [U]). Myocardial Heterogeneity Index (Hi) was measured by an automated analysis developed in our research unit. Hi was finally calculated from images SPECT using a Markovian analysis. For this study Hi is given by the equation: Hi = Σm [1/(1+m)2]Pd(m).

SECONDARY OUTCOMES:
scintigraphy | day 0 (inclusion)
  An FFR value of 0.80 or less identifies ischemia-causing coronary stenoses. The global summed stress score (SSS) was calculated by adding the scores of the 17 segments in the stress and rest images, respectively. Scans were considered as normal when SSS was < 4.

CONTACTS AND LOCATIONS:
Overall Officials: BARONE ROCHETTE MD Gilles, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, Isère, France